CLINICAL TRIAL: NCT00890721
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Single Administration of SKY0402 for Prolonged Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy
Brief Title: Study of Pain Control in Hemorrhoidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402C316
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Hemorrhoid
Keywords: Hemorrhoid; Hemorrhoidectomy; Postoperative pain; Analgesia
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative; Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKY0402 (Experimental): During the hemorrhoidectomy, 30cc of SKY0402 is injected into the wound.
  Interventions: Drug: SKY0402
- Placebo (Placebo Comparator): During the hemorrhoidectomy, 30cc Placebo injected into the wound.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKY0402 — During the operation, 30cc of SKY0402 are injected into the wound.
  Other Names: EXPAREL
  Arms: SKY0402
Drug: Placebo — During the hemorrhoidectomy, 30cc Placebo injected into the wound.
  Other Names: saline 0.9%
  Arms: Placebo

SUMMARY:
Patients will get an injection of either SKY0402 or placebo during hemorrhoid surgery, and their pain and pain medicine use will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age at the Screening visit
* American Society of Anesthesiologists (ASA) class 1-3
* Scheduled to have a two or three column excisional hemorrhoidectomy under general anesthesia using the Milligan-Morgan technique
* For female subjects, surgically sterile or at least two years menopausal, or using an acceptable method of birth control; must have a documented negative blood or urine pregnancy test within 24 hours before surgery
* Clinical lab values less than or equal to twice the upper limit of normal or, if abnormal, deemed not clinically significant per the Investigator.
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments
* Able to speak, read, and understand the language of all subject-facing documents, including the ICF and study questionnaires
* Able and willing to comply with all study visits and procedures

Exclusion Criteria:

* Single-column hemorrhoidectomy or hemorrhoidectomy without an internal component
* Body weight less than 50 kilograms (110 pounds)
* History of hypersensitivity or idiosyncratic reactions or amide-type local anesthetics, opioids, or propofol
* Current painful physical condition or concurrent surgery other than hemorrhoids that may require analgesic treatment (such as non-steroidal anti-inflammatory drug [NSAID], opioid, selective serotonin reuptake inhibitor [SSRI], tricyclic antidepressant, gabapentin, pregabalin) in the postoperative period for pain that is not strictly related to the hemorrhoidectomy procedure and may confound the postoperative assessments
* Concurrent fissurectomy
* Use of any NSAID including selective COX-2 inhibitor, opioid, SSRI, tricyclic antidepressant, gabapentin, or pregabalin within three days of surgery
* Use of acetaminophen within 24 hours of surgery
* Chronic users of analgesic medications, including taking opioid medications for more than 14 days in the last 3 months, or non-opioid pain medications more than 5 times per week
* History of, suspected, or known addiction to or abuse of drugs or alcohol within the past two years
* Current use of glucocorticosteroids or use of glucocorticoids within one month of enrollment into this study
* HIV infection or hepatitis
* Currently pregnant, nursing, or planning to become pregnant during the course of the study or within one month of study drug administration
* Any psychiatric, psychological, medical, or laboratory condition that the investigator feels makes the subject an inappropriate candidate for this clinical trial
* Subjects who have received another investigational drug within the longer of the last 30 days or 10 elimination half-lives
* Previous participation in a SKY0402 study
* Failure to pass drug and alcohol screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Śledziński, MD, Principal Investigator — General Surgery, Transplantology and Endocrinology Department, Gdansk
Locations (1):
- Prof. Zbigniew Śledziński, Gdansk, Poland

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SKY0402 | Placebo
Started | 95 | 94
Completed | 94 | 93
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SKY0402 | Placebo | Total
Number analyzed (Participants) | 95 | 94 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 86 | 172
  >=65 years | 9 | 8 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (12.2) | 48.7 (12) | 48.4 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 63 | 67 | 130
Region of Enrollment [Number; unit: participants]
  Poland | 36 | 36 | 72
  Serbia | 25 | 25 | 50
  Georgia | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Curve (AUC) of the Numeric Rating Scale at Rest (NRS-R) Pain Intensity Scores Through 72 Hours for Subjects Receiving SKY0402 vs. Placebo.
Description: To assess pain intensity at rest (NRS-R), the subject was to assume a resting position that did not exacerbate his or her postoperative pain and respond to the following question: "On a scale of 0 to 10, where 0 = no pain and 10 = worst possible pain, how much pain are you having right now?"
Time Frame: 72 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hr
Arm/Group | SKY0402 | Placebo
Number analyzed (Participants) | 94 | 93
units on a scale*hr | 141.8 (10.7) | 202.5 (10.7)

2. Secondary Outcome: Participants With Adverse Events Through 72 Hours or Serious Adverse Events Through 30 Days
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SKY0402 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/94 | 1/93
Other Adverse Events (participants affected / at risk) | 2/94 | 5/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SKY0402 (N=94) | Placebo (N=93)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SKY0402 (N=94) | Placebo (N=93)
Painful defaecation (Gastrointestinal disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No